CLINICAL TRIAL: NCT00074607
Title: Intrathecal Gemcitabine Therapy for Neoplastic Meningitis: A Phase I and Pharmacokinetic Study
Brief Title: Intrathecal Gemcitabine to Treat Neoplastic Meningitis, IT Gemcitabine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Pittsburgh (Other); National Cancer Institute (NCI) (NIH); Children's Hospital of Pittsburg (Unknown); Seattle Children's Hospital (Other); Mayo Clinic (Other); Brown University (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor of Pediatrics-Hem-Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10564 IT Gemcitabine; I.T. Gemcitabine (Other: Baylor College of Medicine); NCT00039143 (obsolete NCT alias); NCT00048243 (obsolete NCT alias); NCT00052806 (obsolete NCT alias)
Record Dates: First submitted 2003-12-16; First posted 2003-12-18 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Meningitis; Neoplasms
Keywords: Neoplastic meningitis
MeSH Terms: conditions — Meningitis; Neoplasms; Meningeal Carcinomatosis | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrathecal gemcitabine administration (Experimental): Intrathecal gemcitabine will be given on a weekly schedule for the first cohort of patients at the 5 mg dose level and then a twice-weekly (i.e., every 3 to 4 days) schedule. Drug administration will be by the intraventricular (Ommaya reservoir injection) route.
  Patients will be hospitalized overnight following their first dose of gemcitabine. If the first dose is well tolerated, subsequent induction doses may be administered in the outpatient setting with close observation for a minimum of 2 hours after administration.
  Dose Levels and Dose Escalation:
  Dose Level 1a: 5 mg
  Dose Level 1b: 5 mg
  Dose Level 2: 10 mg
  Dose Level 3: 20 mg
  Dose Level 4: 30 mg
  Dose Level 5: 40 mg
  Dose Level 6: 50 mg
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Schedule
  Induction: At Dose Level 1athe first cohort of patients will receive intrathecal gemcitabine on a weekly basis for a total of 6 weeks. If that is tolerated, the subsequent cohort will receive intrathecal gemcitabine on a twice-weekly basis (Dose Level 1b) for a total of 6 weeks. Subsequent cohorts (Dose Levels 2 - 6) will receive intrathecal gemcitabine on a twice weekly basis for a total of 6 weeks (12 doses).
  In the absence of disease progression or DLT, patients may proceed to consolidation.
  Consolidation: Intrathecal gemcitabine will be administered weekly for a total of 6 doses. The first dose of consolidation will be given 1 week after the last induction dose. In the absence of disease progression or DLT, patients may proceed to maintenance.
  Maintenance: Intrathecal gemcitabine will be given twice monthly for 4 months and monthly thereafter. In the absence of progressive disease or dose-limiting toxicity, the total duration of therapy will be 1 year.
  Other Names: Gemzar

SUMMARY:
Subject's are being asked to take part in this study because he or she has a type of cancer that has spread to the meninges (tissues that cover the brain and spinal cord).

There is no known effective treatment for this specific disease or the subject has received all of the treatments that are known to work for his or her specific disease without success. Currently, there is no other effective treatment for this type of cancer.

The purposes of this study are:

* to determine the highest dose of gemcitabine, an anti-cancer drug, that can safely be given directly into the spinal fluid of children and adults whose cancer no longer responds to standard treatment;
* to find out what effects (good and bad) gemcitabine has when given directly into the cerebrospinal fluid (called intrathecal administration) in children and adults with neoplastic meningitis (cancer that has spread to the lining of the brain and spinal cord);
* to determine if gemcitabine is beneficial to the patient;
* to understand how gemcitabine is handled by the body after intrathecal administration.

DETAILED DESCRIPTION:
WHAT IS INVOLVED IN THE STUDY? Before participating in this study, there will be a screening process.

Administration:

Gemcitabine will be received directly into the cerebrospinal fluid (fluid that circulates around the brain and spinal cord) through an Ommaya reservoir (or other similar type of reservoir). An Ommaya reservoir is a surgically implanted catheter that is used to inject medication or to withdraw cerebrospinal fluid from the fluid chambers in the head.

All patients will be hospitalized overnight following their first dose of gemcitabine. If the first dose is well tolerated, further doses of gemcitabine will be administered in the outpatient clinic with close observation for a minimum of 2 hours after administration.

Weeks 1-6 Cohort 1a (first three patients):

Gemcitabine will be given once a week for 6 weeks. Patients may continue therapy if the disease has not worsened.

Weeks 1-6 (all other patients enrolled on this study):

Gemcitabine will be given twice a week for 6 weeks. Patients may continue therapy if the disease has not worsened.

Weeks 7-12:

Gemcitabine will be given once a week for 6 weeks.

Weeks 13-29 (approximately):

Gemcitabine will be given twice monthly for 4 months.

Weeks 30-52 (approximately):

Gemcitabine will be given monthly for the duration of the study.

For safety reasons, the first patients treated in the study will receive a low dose of gemcitabine. If that dose does not cause severe side effects, the next group will receive a higher dose of gemcitabine than given to the earlier group, or may receive a lower dose if side effects occur. In addition, the first three patients treated on this study will receive the gemcitabine once weekly. If this is tolerated, subsequent patients will receive the medication twice weekly.

Following the first dose of gemcitabine investigators would like to draw special blood and spinal fluid samples to help learn how much of the drug is in the blood and spinal fluid. These studies are called pharmacokinetics. A total of 10 samples will be collected. The blood samples may be collected from an intravenous catheter or a central venous catheter. The spinal fluid samples may be collected either via Ommaya reservoir or lumbar reservoir.

In addition to intrathecal gemcitabine, the patient may receive other chemotherapy, not given directly into the fluid surrounding the brain and spine, as recommended by his or her doctor for the treatment or prevention of cancer outside the lining of the brain and spinal cord.

The maximum length of treatment with gemcitabine is one year. However, at the end of the study, monthly check-ups are required to monitor the disease and to make sure that any side effects from the study drug have stopped.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 years of age.
* Neoplastic meningitis secondary to an underlying leukemia/lymphoma or a solid tumor (including primary CNS tumors or carcinomas of unknown primary site) for which there is no conventional therapy. Patients with CNS leukemia/lymphoma must be refractory to conventional therapy, including XRT (i.e. 2nd or greater relapse). Neoplastic meningitis is defined as follows:

  * Leukemia/Lymphoma: CSF cell count > 5 uL AND evidence of blast cells on cytospin preparation or by cytology.
  * Solid tumor: Presence of tumor cells on cytospin preparation or cytology OR presence of meningeal disease on MRI scans.
* Life expectancy of at least 6 weeks.
* Patients > 10 years old: Karnofsky performance status of >/= 50%. Patients </=10 years old: Lansky performance status of >/= 50%.
* Must have recovered from the acute neurotoxic effects of all prior chemo, immuno, or radiotherapy and must be without uncontrolled significant systemic illness (e.g. infection). Must not have received any systemic CNS-directed therapy within 3 weeks or craniospinal irradiation within 8 weeks prior to starting treatment on study. Must not have received any intrathecal therapy within 1 week prior to starting treatment on study.
* Must have a platelet count >40,000/uL and HCT >30% and an ANC of > 1000/uL.
* Must have adequate liver function, total bilirubin < 2.0 mg, SGPT < 5 times upper limits of normal; adequate renal function (serum creatinine < 2 times upper limits of normal for age).
* Patients must have or be willing to have an intraventricular access device such as an Ommaya reservoir.

Exclusion Criteria:

* Patients receiving other therapy (either intrathecal or systemic) designed to treat their leptomeningeal disease. However, patients receiving concomitant chemotherapy to control systemic disease or bulk CNS disease will be eligible, provided that the systemic chemotherapy is not a phase I agent, an agent that significantly penetrates the CSF, or an agent known to have serious unpredictable CNS side effects.
* Nuclear Medicine CSF flow studies are required within the 2 weeks prior to study entry for all solid tumor patients. In leukemia/lymphoma patients a CSF flow study is only required if CSF analysis or an MRI suggests that there is a blockage to CSF flow. Patients with clinical evidence of obstructive hydrocephalus are not eligible for this protocol. Nor are patients with compartmentalization of CSF flow as documented by radioisotope Indium111 or Technetium99-DTPA flow eligible for this protocol. If a CSF flow block or compartmentalization is demonstrated, focal radiotherapy to the site of the block to restore flow followed by a repeat CSF flow study demonstrating clearing of the blockage is required for the patient to be eligible for the study.
* Patients must not have clinically significant abnormalities of serum electrolytes, including calcium, magnesium, and phosphorus.
* Patients with a ventriculoperitoneal (VP) or ventriculoatrial (VA) shunt are not eligible unless they are shunt-independent and there is evidence that their shunt is nonfunctional
* Patients who have leukemia/lymphoma with a concomitant bone marrow relapse.
* Women of childbearing age must not be pregnant or lactating. (Male and female patients who are fertile must be willing to use an effective means of birth control to avoid pregnancy.)
* Must be free of uncontrolled infection except HIV (i.e., AIDS-related lymphomatous meningitis).
* Must NOT be receiving any other investigational agents and must not have received any other investigational agent within 14 days prior to study treatment. The 14-day period should be extended if the investigational agent is known to have delayed toxicity.
* Patients with impending spinal cord compression, CNS involvement requiring local XRT (e.g. optic nerve), or isolated bulky ventricular or leptomeningeal based lesions are not eligible.
* Concomitant CNS radiation therapy is not permitted. (Patients are not permitted to receive radiation to any port that encompasses any part of the brain or spine while on study.) Patients may receive radiation therapy to extra-CNS sites, e.g. painful bone metastases not in the craniospinal axis.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-12; Primary Completion 2005-07 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Asses the toxicity of intrathecally administered gemcitabine in a limited dosage escalation schedule. | 1 year
Determination of the maximum tolerated dose of intrathecally administered gemcitabine. | 4 weeks
  The MTD of IT gemcitabine will be that dose at which less than 20% of patients experience DLT as defined earlier. Escalations are planned in groups of three patients, with an additional three patients to be added at the first indication of DLT.

SECONDARY OUTCOMES:
To define the plasma and CSF pharmacokinetics of gemcitabine and its major metabolite, 2', 2'-difluoro-deoxyuridine (dFdU) after intrathecal administration. | 1 year
Documentation of any responses following intrathecal gemcitabine administration. | 1 year
Investigate MMP expression in pediatric and adult patients with a variety of primary diseases. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - National Cancer Institute, Bethesda, Maryland
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Bernardi RJ, Bomgaars L, Fox E, Balis FM, Egorin MJ, Lagattuta TF, Aikin A, Whitcomb P, Renbarger J, Lieberman FS, Berg SL, Blaney SM. Phase I clinical trial of intrathecal gemcitabine in patients with neoplastic meningitis. Cancer Chemother Pharmacol. 2008 Jul;62(2):355-61. doi: 10.1007/s00280-007-0601-x. Epub 2007 Oct 2. PMID 17909804